CLINICAL TRIAL: NCT05757869
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy, Parallel Group, Active-Controlled Study to Evaluate the Efficacy and Safety of Milvexian, an Oral Factor XIa Inhibitor, Versus Apixaban in Participants With Atrial Fibrillation
Brief Title: A Study of Milvexian Versus Apixaban in Participants With Atrial Fibrillation
Acronym: LIBREXIA-AF
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109220; 70033093AFL3002 (Other: Janssen Research & Development, LLC); 2022-501419-15-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — milvexian; apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Milvexian (Experimental): Participants will receive milvexian 100 milligrams (mg) orally, twice daily and placebo that matches apixaban beginning on Day 1 through end of treatment (EOT). Participants after the EOT visit may have an option to receive open-label apixaban at the appropriate dose (5 mg or 2.5 mg, twice daily), for which the sponsor provides a 30-day supply.
  Interventions: Drug: Milvexian; Drug: Placebo
- Apixaban (Active Comparator): Participants will receive a placebo that matches milvexian and a capsule containing apixaban 5 mg or 2.5 mg orally, twice daily. Participants after the EOT visit may have an option to receive open-label apixaban (5 mg or 2.5 mg, twice daily) at the appropriate dose, for which the sponsor provides a 30-day supply.
  Interventions: Drug: Apixaban; Drug: Apixaban Placebo

INTERVENTIONS:
Drug: Milvexian — Milvexian will be administered orally.
  Arms: Milvexian
Drug: Apixaban — Apixaban will be administered orally.
  Arms: Apixaban
Drug: Placebo — Milvexian matching milvexian placebo will be administered orally.
  Arms: Milvexian
Drug: Apixaban Placebo — Apixaban matching apixaban placebo will be administered orally.
  Arms: Apixaban

SUMMARY:
The purpose of this study is to evaluate if milvexian is at least as effective as apixaban for reducing the risk of the composite stroke and non-central nervous system (CNS) systemic embolism.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Medically stable and appropriate for chronic antithrombotic treatment
* Atrial fibrillation eligible to receive anticoagulation
* Participant must satisfy one or both of the following categories of risk factors (a or b): a) one or more of the following risk factors: i) age greater than or equal to 75 years, ii) history of any type of stroke including symptomatic stroke of any kind. b) two or more of the following risk factors: i) age between 65 and 74 years, ii) hypertension, iii) diabetes mellitus, iv) atherosclerotic vascular disease, v) heart failure

Exclusion Criteria:

* Hemodynamically significant valve disease or those with valve disease that will potentially require surgical valve replacement during the study
* Any condition other than AF that requires chronic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20283 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to the First Occurrence of Composite Endpoint of Stroke and Non-central nervous system (CNS) Systemic Embolism | Up to 4 years
  Time to the first occurrence of composite endpoint of stroke and non-CNS systemic embolism will be reported.

SECONDARY OUTCOMES:
Time to the First Occurrence of International Society of Thrombosis and Hemostasis (ISTH) Major Bleeding | Up to 4 years
  Time to the first occurrence of ISTH major bleeding will be reported.
Time to the First Occurrence of the Composite of ISTH Major and Clinically Relevant Non-major (CRNM) Bleeding | Up to 4 years
  Time to the first occurrence of the composite of ISTH major and CRNM bleeding will be reported.
Time to the First Occurrence of Composite Endpoint of Stroke, Non-CNS Systemic Embolism and ISTH Major Bleeding | Up to 4 years
  Time to the first occurrence of composite endpoint of stroke, non-CNS systemic embolism and ISTH major bleeding will be reported.
Time to the First Occurrence of Composite Endpoint of Cardiovascular (CV) Death, Myocardial Infarction (MI), Stroke, and Non-CNS Systemic Embolism | Up to 4 years
  Time to the first occurrence of composite endpoint of CV death, MI, stroke, and non-CNS systemic embolism will be reported.
Time to CV Death | Up to 4 years
  Time to CV death will be reported.
Time to the First Occurrence of Composite Endpoint of All-cause Death, MI, Stroke and Non-CNS Systemic Embolism | Up to 4 years
  Time to the first occurrence of composite endpoint of all-cause death, MI, stroke and Non-CNS systemic embolism will be reported.
Time to the First Occurrence of Composite Endpoint of CV Death, MI, Stroke, Acute Limb Ischemia (ALI), and Urgent Hospitalization for Vascular cause of Ischemic Nature | Up to 4 years
  Time to the first occurrence of composite endpoint of CV death, MI, stroke, ALI [any unanticipated revascularization or amputation of ischemic limb]), and urgent hospitalization for vascular cause of ischemic nature (including deep vein thrombosis [DVT] and pulmonary embolism [PE]) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1038):
- United States (214):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - Ascension St. Vincent's Health System, Birmingham, Alabama
  - SEC Clinical Research, Dothan, Alabama
  - HH Heart Center and Heart Center, Huntsville, Alabama
  - CB Flock Research Corporation, Mobile, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Valleywise Health Medical Center, Phoenix, Arizona
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Arizona Heart Hospital, Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Vitality Clinical Research, Beverly Hills, California
  - Chula Vista Cardiac Clinic, Chula Vista, California
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Mission Cardiovascular Research Institute, Fremont, California
  - Paradise Clinical Research Group LLC, Glendora, California
  - Miller Children's at Long Beach Medical Center, Long Beach, California
  - Los Angeles Cardiology Associates, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Merced Vein and Vascular Center, Merced, California
  - Radin Cardiovascular Medical Group, Newport Beach, California
  - California Medical Research Associates, Inc., Northridge, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Health Care, Palm Springs, California
  - Havana Research Institute LLC, Pasadena, California
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - Stanford Health Care, Redwood City, California
  - San Diego Cardiac Center, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Ramin Manshadi, MD, Stockton, California
  - UCLA School of Medicine, Torrance, California
  - Cardiology Associates Medical Group, Ventura, California
  - North County Internal Medicine, Vista, California
  - John Muir Physician Network Clin. Research Center, Walnut Creek, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - Paradigm Clinical Research Centers, Inc., Wheat Ridge, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Western Connecticut Health Network/Danbury Hospital, Danbury, Connecticut
  - Cardiology Associates of Fairfield County, Stamford, Connecticut
  - PriMed Physicians, A Member of NE Medical Group, Trumbull, Connecticut
  - Cardiology Physicians, Newark, Delaware
  - George Washington University School of Medicine, Washington D.C., District of Columbia
  - Orlando Heart Specialists, Altamonte Springs, Florida
  - Bay Area Cardiology Associates, P.A. - Brandon Office, Brandon, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Cardiology Consultants, Daytona Beach, Florida
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - Accel Research Sites, DeLand, Florida
  - The Cardiac & Vascular Institute Research Foundation, Gainesville, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Clearwater Cardiovascular Consultants, Largo, Florida
  - Miami Clinical Research, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Ascension Sacred Heart Hospital, Miramar Beach, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Central Florida Medical Associates, Orange City, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Cardiology Consultants, Pensacola, Florida
  - North Broward Hospital District, Pompano Beach, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Coastal Cardiology Consultants, Safety Harbor, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Adtremed Inc, Tampa, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - Helping Hands Health Center dba Helping Hands Evolution Research, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Atlanta Heart Specialists, Cumming, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Cardiology Consultants of South Georgia Inc, Thomasville, Georgia
  - The Queens Medical Center, Honolulu, Hawaii
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Clinical Investigation Specialists, Gurnee, Illinois
  - Chicago Medical Research, LLC, Hazel Crest, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Prairie Education And Research Cooperative, O'Fallon, Illinois
  - Advocate Heart Institute, Oak Lawn, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Blessing Hospital, Quincy, Illinois
  - OSF HealthCare Cardiovascular Institute, Rockford, Illinois
  - Springfield Clinic 1st, Springfield, Illinois
  - Bloomington Hospital, Bloomington, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - St. Elizabeth Physicians, Crittenden, Kentucky
  - Kentuckyone Health Neurology Associates, Louisville, Kentucky
  - Owensboro Medical Practice, Owensboro, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Grace Research, LLC - Bossier City, Bossier City, Louisiana
  - Medical Research Specialists, Chalmette, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Pierremont Cardiology, Shreveport, Louisiana
  - Clinical Trials of America, West Monroe, Louisiana
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Shady Grove Office, Rockville, Maryland
  - Tidal Health Peninsula Regional Inc., Salisbury, Maryland
  - Spectrum Clinical Research, Inc., Towson, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Flint Clinical Research, Flint, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan Heart & Vascular Institute, Petoskey, Michigan
  - Revival Research Institute LLC, Southgate, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Trinity Health Michigan d b a Michigan Heart, Ypsilanti, Michigan
  - HealthPartners Institute, Bloomington, Minnesota
  - Essentia Health SMDC, Duluth, Minnesota
  - Fairview Health System, Maplewood, Minnesota
  - Mississippi Baptist Health Systems, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - The Curators of the University of Missouri on behalf of University of Missouri Health Care, Columbia, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Virtua Medical Group, PA, Marlton, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - NYU Hudson Valley Cardiology, Cortlandt Manor, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Westchester Medical Center Advanced Physician Services PC, Kingston, New York
  - Laurelton Heart Specialist, PC, Laurelton, New York
  - Crystal Run Healthcare LLP, Middletown, New York
  - NYU Langone Hospital Long Island, Mineola, New York
  - Weill Cornell Medical College, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Cardiac Care & Vascular Medicine, PLLC, The Bronx, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Clinical Trials of America, Lenoir, North Carolina
  - Pinehurst Medical Clinic Inc, Pinehurst, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Trinity Medical Group, Minot, North Dakota
  - Summa Health System, Akron, Ohio
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Louis Stokes Cleveland VA Med Ctr, Cleveland, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Dayton Heart Center, Dayton, Ohio
  - Advanced Medical Research, Maumee, Ohio
  - The Heart House, Springfield, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Ascension Medical Group - St. John Clinic Infectious Disease, Bartlesville, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - St John Health System Inc, Tulsa, Oklahoma
  - Providence Heart Clinic, Portland, Oregon
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Hamot Medical Center, Erie, Pennsylvania
  - Capital Area Research, Newport, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Hudson Valley Cardiovascular Practice, PC, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation, Sayre, Pennsylvania
  - Geisinger Medical Center, Scranton, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - York Hospital, York, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Internal Medicine Associates of Anderson, Anderson, South Carolina
  - MUSC Health Heart Vascular Columbia Medical Park DT III, Columbia, South Carolina
  - St. Francis Physician Services, Inc, DBA Upstate Cardiology Research, Greenville, South Carolina
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Jackson Clinic, Jackson, Tennessee
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Wellmont CVA Heart Institute, Johnson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - East Tennessee Heart Consultants, Knoxville, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Cardiovascular Associates, Powell, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Amarillo Heart Clinical Research Institute, Amarillo, Texas
  - Ascension Texas Cardiovascular, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Texas Health Dallas, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - East Texas Cardiology, PA, Houston, Texas
  - Primecare Medical Group, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Novel Research LLC, Houston, Texas
  - West Houston Area Clinical Trial Consultants LLC, Katy, Texas
  - Texas Cardiology Research Center, Kingwood, Texas
  - Odessa Heart Institute, Odessa, Texas
  - Sun Research Institute, San Antonio, Texas
  - Southwest Medical Clinic, Sugar Land, Texas
  - Northwest Houston Clinical Research, Tomball, Texas
  - Baylor Scott and White Research Institute, Waco, Texas
  - Alpine Research Organization, Farmington, Utah
  - Burke Internal Medicine and Research, Burke, Virginia
  - Roanoke Heart Institute PLC, Roanoke, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
  - Universal Research Group, LLC, Tacoma, Washington
  - Wausau Hospital, Wausau, Wisconsin
  - Allegiance Reserach Specialists, LLC, Wauwatosa, Wisconsin
- Argentina (50):
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca
  - CEDIC Centro de Investigaciones Clinicas, Buenos Aires
  - CIPREC, Buenos Aires
  - Sanatorio Finochietto, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - CEMEDIC, Buenos Aires
  - CINME Centro de Investigaciones Metabolicas, CABA
  - Clínica y Maternidad Suizo Argentina, Capital Federal
  - Consultorio Dr. Litvak Bruno, Ciudad Autonoma Buenos Aires
  - Consultorios Asociados de Endocrinología e Investigación Clínica Aplicada, Ciudad Autonoma Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - Glenny Corp. S.A. - Bioclinica Argentina, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad de Buenos Aires
  - Instituto Médico Elsa Pérez I.M.E.P, Ciudadela
  - Centro Médico Colón, Cordooba
  - Clinica Coronel Suarez, Coronel Suárez
  - Clinica Privada Velez Sarsfield, Córdoba
  - Clínica Colombo, Córdoba
  - Hospital San Roque, Córdoba
  - Instituto Privado de Investigaciones Clinicas de Cordoba, Córdoba
  - CIDIM-Centro Integral de Diagnostico por Imagenes Marchegiani, Córdoba
  - Sanatorio Allende, Córdoba
  - Instituto Privado De Especialidades Medicas S.A. Fundacion J Robert Cade, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Hospital Italiano de Cordoba, Córdoba
  - Hospital Cordoba, Córdoba
  - Centro Medico Luquez, Córdoba
  - CIPADI, Godoy Cruz
  - Centro Medico Lebensohn, Junín
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes
  - DIM Clinica Privada, Ramos Mejía
  - Sanatorio Britanico S.A., Rosario
  - Sanatorio de la Mujer, Rosario
  - Instituto de Investigaciones Clinicas de Rosario, Rosario
  - Sanatorio Parque, Rosario
  - Centro de Investigaciones Clinicas Salta, Salta
  - Centro Cardiovascular Salta, Salta
  - Investigaciones Clinicas Cuyo, San Juan
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Instituto de Investigaciones Clinicas San Nicolas, San Nicolás
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Hospital Provincial Dr. Jose Maria Cullen, Santa Fe
  - Centro de Investigaciones Médicas Temperley, Temperley
  - Sanatorio San Martin, Venado Tuerto
  - Clinica Privada Fusavim SRL, Villa María
  - Instituto de Investigaciones Clínicas Zarate, Zárate
- Australia (12):
  - Flinders Medical Centre, Adelaide
  - Advara HeartCare Wesley, Brisbane
  - Concord Repatriation General Hospital, Concord
  - Peninsula Heart Center, Frankston
  - The Canberra Hospital, Garran
  - Royal Brisbane and Women's Hospital, Herston
  - GenesisCare Joondalup-Shenton House, Joondalup
  - Novatrials, Kotara
  - GenesisCare, Leabrook
  - Liverpool Hospital, Liverpool
  - Core Research Group, Milton
  - Brisbane Health Connect, Tarragindi
- Belgium (14):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
  - CSL Arlon, Arlon
  - C.H.U. Brugmann, Brussels
  - CUB Hôpital Erasme, Brussels
  - AZ Sint-Blasius, Dendermonde
  - UZA, Edegem
  - Jessa Ziekenhuis - Campus St.-Ursula, Herk-de-Stad
  - Chu Tivoli, La Louvière
  - UZ Leuven, Leuven
  - Az Sint-Maarten, Mechelen
  - Heilig Hart Ziekenhuis Lier, Mol
  - AZ Delta VZW, Roeselare
  - AZ Turnhout, Turnhout
- Brazil (45):
  - Hospital Felício Rocho, Belo Horizonte
  - Hospital Vera Cruz, Belo Horizonte
  - Cardresearch - Cardiologia Assistencial, Belo Horizonte
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Rede D or Sao Luiz S A Hospital do Coracao do Brasil, Brasília
  - Centro de Cardiologia Clinica e Pesquisa Doutora Juliana Souza Ltda CECAP Centro de Cardiologia Clinica, Brasília
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul
  - C.E.C.-Centro Especializado em Cardiologia Ltda.- Loema Medicina e Bem Estar, Campinas
  - Instituto de Pesquisa Clinica de Campinas, Campinas
  - Hospital Universitario, Canoas
  - Sociedade Literaria e Caritativa Santo Agostinho Hospital Sao Jose, Criciúma
  - Irmandade Santa Casa de Misericórdia de Curitiba -Pontifícia Universidade Católica do Paraná-PUCPR, Curitiba
  - Hospital Cardiológico Costantini, Curitiba
  - Núcleo de Pesquisa Clinica, Curitiba
  - Universidade Federal de Goias - Hospital das Clinicas da UFG, Goiânia
  - Instituto do Coracao de Marília, Marília
  - Irmandade da Santa Casa de Misericórdia de Marília, Marília
  - Hemocardio SS Ltda, Natal
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Santa Casa de Misericordia de Pelotas, Pelotas
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - IMV Pesquisa Cardiologica Sociedade Simples HMD COR l, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - Fundacao Universitaria de Cardiologia, Porto Alegre
  - Pro Cardiaco Pronto Socorro Cardiologico, Recife
  - Secretaria de Saude Hospital Agamenon Magalhaes, Recife
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Impar Servicos Hospitalares S/A, Rio de Janeiro
  - Instituto CardioPulmonar, Salvador
  - Fundacao Bahiana de Cardiologia, Salvador
  - Pesquisare Saude, Santo André
  - Instituto de Cardiologia de Santa Catarina, São José
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - FGM Clinica Paulista de Doencas Cardiovasculares Ltda IPDC Cardiologia, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
  - Instituto de Moléstias Cardiovasculares Tatuí, Tatuí
  - HC-UFTM - Hospital de Clínicas da Universidade Federal do Triângulo Mineiro, Uberaba
  - Clinica Cardioped Ltda, Vitória
  - CEDOES, Vitória
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga
- Bulgaria (38):
  - MHAT Puls, Blagoevgrad
  - MC 4Life Ltd, Burgas
  - Medical Center Diamedical, Dimitrovgrad
  - MHAT St. Ekaterina, Dimitrovgrad
  - Medical Centre Asklepii OOD, Dupnitsa
  - Multiprofile Hospital for Active Treatment Dr. Tota Venkova, Gabrovo
  - Multiprofile Hospital for Active Treatment - Haskovo, Haskovo
  - Medical center Rodopimed EOOD, Kardzhali
  - UMHAT 'Pulmed' OOD- MS 'Zdrave' - Pazardzhik, Pazardzhik
  - Exacta Medica, Pleven
  - Medical Center Medconsult-Pleven, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT 'Heart and Brain Center for Excellence', Pleven
  - UMHAT 'Sv. Georgi' EAD, Plovdiv
  - Medical Center- Prolet Ltd, Rousse
  - MC Rusemed ltd, Rousse
  - Medical Center Unimed Eood, Sevlievo
  - Individual Ambulatory of Cardiology, Sofia
  - DCC Ascendent EAD, Sofia
  - Second Multiprofile Hospital for Active Treatment MHAT - Sofia AD, Sofia
  - MHAT Knyaginya Klementina, Sofia
  - National Multiprofile Transport Hospital Tsar Boris III, Sofia
  - Multiprofile Hospital For Active Treatment National Cardiology Hospital, Ead, Sofia
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - Diagnostic Consultation Centre 'Alexandrovska' EOOD, Sofia
  - UMHAT Prof. Dr. Aleksandar Chirkov, Sofia
  - Medical Center Hera EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment - Tsaritsa Yoanna - ISUL, EAD, Sofia
  - Meditsinski Centar - Izgrev Eood, Sofia
  - DCC Convex EOOD, Sofia
  - Medical Centre Kalimat, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
  - Medical Center ZaraMed, Stara Zagora
  - UMHAT Prof. Dr. St. Kirkovich AD, Stara Zagora
  - DCC Chaika EOOD, Varna
  - Medical Center -Medika Plus, Veliko Tarnovo
  - MHAT Dr Stefan Cherkezov, Veliko Tarnovo
  - MHAT Sv. Panteleymon AD, Yambol
- Canada (16):
  - The Governers of the University of Calgary, Calgery, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Victoria Cardiac Arrhythmia Trials Inc, Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Brampton Research Assoc, Brampton, Ontario
  - Dr. Saul Vizel Cardiac Research Office, Cambridge, Ontario
  - One Heart Care, Mississauga, Ontario
  - Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - CPS Research, Waterloo, Ontario
  - ViaCar Recherche Clinique Inc, Greenfield Park, Quebec
  - CHUM - Pavillon B, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Montreal Heart Institute, Québec, Quebec
- Chile (10):
  - Quantum Research, Puerto Varas
  - Enroll Spa, Santiago
  - BioMedica Research Group, Santiago
  - SMOLAM, Santiago
  - Centro de Investigacion Clinica Universidad Catolica de Chile CICUC, Santiago
  - CeCim - Centro de Estudios Clinicos e Investigacion Medica, Santiago
  - Sociedad Medica Cardiologica El Llano, Santiago
  - Centro de Estudios Cardiologicos y de Medicina Interna, Temuco
  - Centro de Investigacion Clinica del Sur, Temuco
  - Centro de Estudios Clinicos V Region Ltda, Viña del Mar
- China (66):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Cangzhou People's Hospital, Cangzhou
  - Jilin Province Peoples Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital of Central South University, Changsha
  - The Third Hospital of Changsha, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Chongqing General Hospital, Chongqing
  - Heilongjiang Daqing People's Hospital, Daqing
  - Dongguan People s Hospital, Dongguan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Jiangxi Ganzhou Peoples Hospital, Ganzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - ZhuJiang Hospital of Southern Medical University, Guangzhou
  - The Third Affiliated Hospital Sun Yat sen University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - GuiZhou Privicial Peoples Hospital, Guiyang
  - Affiliated Hospital of Hainan Medical University, Haikou
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou
  - Anhui Province Hospital, Hefei
  - The second hospital of Anhui medical university, Hefei
  - Inner Mongolia People's Hospital, Hohhot
  - Jieyang Peoples Hospital, Jieyang
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Jining No.1 People's Hospital, Jining
  - Lanzhou University Second Hospital, Lanzhou
  - Luoyang Third People's Hospital, Luoyang
  - Jiangxi Provincial Peoples Hospital, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanchang Peoples hospital, Nanchang
  - Ningbo First Hospital, Ningbo
  - Shanghai Ninth Peoples Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Jinshan Hospital Fudan University, Shanghai
  - The First Affiliated Hospital of Shantou University Medical, Shantou
  - Shengjing Hospital Of China Medical University, Shenyang
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Taian City Central Hospital, Taian
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Taizhou First Peoples Hospital, Taizhou
  - Tianjin Chest Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin People's Hospital, Tianjin
  - Tianjin 4th Center Hospital, Tianjin
  - The 2nd Hospital of Tianjin Medical University, Tianjin
  - TEDA International Cardiovascular Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wenzhou Peoples Hospital, Wenzhou
  - The Central Hospital of Wuhan, Wuhan
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Shaanxi Provincial Peoples Hospital, Xi'an
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Northern Jiangsu Peoples Hospital, Yangzhou
  - Yantai Yuhuangding Hospital, Yantai
  - General Hospital of Ningxia Medical Hospital, Yinchuan
  - Affiliated Hospital Of Guangdong Medical University, Zhanjiang
  - The 7th Peoples Hospital of Zhengzhou, Zhengzhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi
- Croatia (10):
  - Zupanijska bolnica Cakovec, Čakovec
  - General Hospital Dubrovnik, Dubrovnik
  - Opća bolnica Karlovac, Karlovac
  - Clinic for Cardiovascular Disease Magdalena, Krapinske Toplice
  - Special Hospital for medical rehabilitation, Krapinske Toplice
  - OB Varazdin, Varaždin
  - Zadar General Hospital, Zadar
  - Poliklinika Solmed, Zagreb
  - Polyclinic Bonifarm, Zagreb
  - University Hospital Dubrava, Zagreb
- Czechia (30):
  - HUMANITAS spol. s r.o., Bílovec
  - MEDICUS SERVICES s.r.o., Brandýs nad Labem
  - Interni ordinace s.r.o, Brandýs nad Labem
  - Vojenska nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - EDUMED s.r.o., Broumov
  - Ordinace pro choroby srdce s.r.o., Chomutov
  - MUDr. Jan Hubac s.r.o., Chrudim
  - Nemocnice Ceske Budejovice a s, České Budějovice
  - Kardiologie KarMa s.r.o, Jablonec nad Nisou
  - Lunacor s.r.o. - Ambulance kardiologie Centrum pro choroby srdce a cev, Kroměříž
  - Kardio Interna s.r.o., Litovel
  - MUDr. Zdenek Vomacka kardiologie a interna s.r.o., Olomouc
  - Fakultni nemocnice Olomouc, Olomouc
  - PreventaMed, s.r.o., Olomouc
  - Cerebrovaskularni poradna s.r.o., Ostrava Poruba
  - Pardubicka krajska nemocnice a s, Pardubice
  - Fakultni nemocnice Plzen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - MUDr. Jan KVASNICKA CSc. Angiologie kardiologie a interna, Prague
  - Nemocnice Na Frantisku, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
  - MUDr. Eva Zídkova, Prague
  - Ustredni vojenske nemocnice Praha, Prague
  - Centrum klinickeho vyzkumu, Příbram
  - Nemocnice Slany, interni oddeleni, Slaný
  - Interni ambulance, Trutnov
  - Interni ambulance Dr.Stanislav Zemek, Uherské Hradiště
  - Cardio Research s r o, Zlín
- Denmark (9):
  - Aarhus University Hospital, Aarhus
  - Amager Hospital, Copenhagen S
  - Gentofte Herlev Hospital, Herlev
  - Herning Regional Hospital, Herning
  - Holbæk Sygehus, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Køge Sygehus Region Sjaelland, Køge
  - Slagelse Sygehus, Slagelse
  - Odense University Hospital, Svendborg
- Dr. Arvo Rosenthal LLC, Tallinn, Estonia
- France (25):
  - CHU Angers - Hopital Hotel Dieu, Angers
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Centre Hospitalier de Beziers, Béziers
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - GH est - Hôpital Cardiovasculaire et Pneumologie Louis Pradel, Bron
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - Hopital Andre Mignot, Le Chesnay
  - CHU de Limoges Hopital Dupuytren, Limoges
  - CHU de la Timone, Marseille
  - Clinique Du Pont De Chaume, Montauban
  - Centre Hospitalier Universitaire - de Nice - Hopital Pasteur, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Broca, Paris
  - Hopital Saint Joseph, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hopital Saint-Antoine, Paris
  - Hopital Cochin, Paris
  - Centre Hospitalier de Pau, Pau
  - Groupe Hospitalier Sud - Hôpital Xavier Arnozan, Pessac
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - CHU Rouen Hopital Charles Nicolle, Rouen
  - Clinique Saint-Hilaire - Centre Frédéric Joliot, Rouen
  - Polyclinique Vauban, Valenciennes
- Germany (45):
  - Klinikum Altenburger Land GmbH, Altenburg
  - Klinikum am Plattenwald, Bad Friedrichshall
  - Kardiologische Praxis Dr. med. univ. Jungmair, Bad Homburg
  - Ruhr Universitat Bochum Diabeteszentrum, Bad Oeynhausen
  - Dres. Haas Kirschner Wagner, Bamberg
  - Vivantes Klinikum Im Friedrichshain, Berlin
  - Augentagesklinik Spreebogen Berlin GbR, Berlin
  - Vivantes Klinikum Am Urban, Abt. fur Kardiologie, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Hellersdorf, Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - GFO Kliniken Bonn, Betriebsstaette St. Marien, Beuel
  - Klinikum Bielefeld, Bielefeld
  - Regiomed Klinikum Coburg, Coburg
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - Gemeinschaftspraxis, Deggingen
  - Praxis-Dr. Frank Menzel, Dessau
  - Stadtisches Klinikum Dresden, Dresden
  - FAZ Dresden-Neustadt GbR, Dresden
  - Hausärztlich-Kardiologisches MVZ Am Felsenkeller GmbH, Dresden
  - ZKS Südbrandenburg GMBH, Elsterwerda
  - Gemeinschaftspraxis Dres. Hagemann und Breiderhoff, Essen
  - Medizentrum Essen Borbeck, Essen
  - Studienzentrum, Essen
  - ClinPhenomics GmbH Co KG Studienzentrum Frankfurt, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - ClinPhenomics GmbH Co KG Studienzentrum Hamburg, Hamburg
  - Praxis Dr. Cornelia Schiewe, Hamburg
  - Medizinisches Versorgungszentrum Prof. Mathey, Prof. Schofer GmbH, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Killat Dr. Holger Kardiologische Praxis, Haßloch
  - Ambulantes Herzzentrum Kassel, Kassel
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Klinikum Ludwigshafen, Ludwigshafen
  - Katholisches Klinikum Mainz; Innere Medizin I- Kardiologie, Mainz
  - Praxis Für Pneumologie Und Allergologie, Mannheim
  - Marienhaus Klinikum, Neuwied
  - GP Dr. Haggenmiller PD Dr. Michael Jeserich, Nuremberg
  - Kardiologische Praxis Papenburg, Papenburg
  - Praxisgemeinschaft Stuhr-Brinkum, Stuhr
  - Universitaetsklinikum Tuebingen, Tübingen
  - Kardiologische Praxis, Wermsdorf
  - Forschungszentrum Ruhr, Witten
  - Stadtkrankenhaus Worms, Worms
  - HELIOS Klinikum Wuppertal GmbH, Wuppertal
- Greece (8):
  - Uni General Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens G Gennimatas, Athens
  - Hippokration Hospital, Athens
  - General Hospital of Nea Ionia 'Konstantopoulio', Athens
  - Onasseio Cardiosurgery Hospital, Kallithea
  - Patras University Hospital, Pátrai
  - Papageorgiou General Hospital, Thessaloniki
  - Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Hungary (35):
  - Lausmed Egeszsegugyi es Szolg. Kft., Baja
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Belgyogyaszati es Kardiologiai Maganrendelo, Békéscsaba
  - Budai Irgalmasrendi Korhaz, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Belvaros-Lipotvaros Egeszsegugyi Szolgalat, Budapest
  - Szt. Rokus Hosp, Budapest
  - Semmelweis Egyetem, Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászati Klinika, Budapest
  - Med-Tima Kft, Budapest
  - Uno Medical Trials Ltd., Budapest
  - Belinus Orvosi es Szamtech. Bt., Debrecen
  - Debreceni Egyetem, Debrecen
  - Bugat Pal Korhaz, Gyöngyös
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - BKS Research Kft, Hatvan
  - Csongrád Megyei Egészségügyi Ellátó Központ Hódmezővásárhely, Hódmezővásárhely
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Bacs-kiskun Megyei Korhaz, Kecskemét
  - Selye Janos Korhaz es Rendelointezet, Komárom
  - IPR Hungary Kft, Miskolc
  - Karolina Korhaz-Rendelointezet, Mosonmagyaróvár
  - TaNaMed Kft., Mosonmagyaróvár
  - Borbanya Praxis Eu. Kft., Nyíregyháza
  - Dr. Nagy Laszlo Kardiologiai Maganrendeles, Orosháza
  - Coromed-Smo Kft, Pécs
  - Szegedi Tudomanyegyetem, Szeged
  - Vita Verum Medical Egeszsegugyi Szolgaltato Bt, Székesfehérvár
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointez, Szolnok
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Belvarosi Egeszseghaz Kft, Zalaegerszeg
  - Obudai Egeszsegugyi Centrum Kft, Zalaegerszeg
- India (28):
  - Jawaharlal Nehru Medical College and Hospital, Aligarh
  - Fortis Escorts Heart Institute and Research Centre, Amritsar
  - Kamal Nayan Bajaj Hospital, Aurangabad
  - St. John's National Academy of Health Sciences - St. John's Medical College Hospital, Bangalore
  - Sri Jayadeva Institute, Bangalore
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre (MRC), Belagavi
  - Bangalore Medical College and Research Institute, Bengaluru
  - S.P.Medical College & AG of Hospitals, Bikaner
  - Tamil Nadu Government Multi Super Speciality Hospital, Chennai
  - S. R. Kalla Memorial General Hospital, Jaipur
  - Eternal Heart Care Centre, Jaipur
  - B M Patel Cardiac Centre, Karamsad
  - Lisie Hospital, Kochi
  - NRS Medical College, Kolkata
  - IPGMER and SSKM Hospital, Kolkata
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - Swasthyam Superspeciality Hospital, Nagar
  - Arneja Heart Institute, Nagpur
  - Central India Cardiology Hospital and Research Institute, Nagpur
  - Chopda Medicare And Research Centre Pvt Ltd Magnum Heart Institute, Nashik
  - All India Institute of Medical Sciences, New Delhi
  - Clinical Research Room, New Delhi
  - Indira Gandhi Institute of Medical Sciences, Patna
  - KEM Hospital & Research Centre, Pune
  - Yashoda Super Speciality Hospitals, Secunderabad
  - Nanjappa Hospital, Shivamogga
  - Government Siddhartha Medical College, Vijayawada
  - King George Hospital, Visakhapatnam
- Israel (14):
  - Haemek Medical Center, Afula
  - Hillel Yaffe Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh Medical Center, Rishon LeZiyyon
  - Ziv Medical Center, Safed
- Italy (26):
  - Ospedale San Donato - ASL 8 Arezzo, Arezzo
  - ASL Caserta_Presidio Ospedaliero San Giuseppe e Melorio_U.O.C. di Cardiologia, Aversa
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Opedaliero-Universitaria Policlinico Sant'orsola Malpighi di Bologna, Bologna
  - AORN Sant'anna e San Sebastiano, Caserta
  - P.O. Vittorio Emanuele Azienda Ospedaliero Universitaria 'Policlinico Vittorio Emanuele', Catania
  - AO di Catanzaro Pugliese Ciaccio, Catanzaro
  - Arcispedale S. Anna Ferrara, Ferrara
  - Ospedale Manzoni, Lecco
  - Fondazione Toscana Gabriele Monasterio CNR, Massa
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - A O Ospedale Niguarda Ca Granda, Milan
  - AOU Policlinico di Modena, Modena
  - Azienda Socio Sanitaria Territoriale di Monza Presidio San Gerardo, Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - AOU Santa Maria della Misericordia di Udine, Perugia
  - A. O.U. Pisana Ospedale di Cisanello, Pisa
  - A.O. San Camillo Forlanini, Roma
  - Ospedale Sandro Pertini di Roma Reparto Emodinamica, Roma
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
  - P.O. Ss. Annunziata, Sassari
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona
- Japan (67):
  - Kasugai Municipal Hospital, Aichi
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Funabashi Municipal Medical Center, Chiba
  - Saiseikai Futsukaichi Hospital, Chikushino-shi
  - Steel Memorial Yawata Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Junshinkai Nakamura Cardiovascular Clinic, Fukuoka
  - Chiba Tokushukai Hospital, Funabashi-shi
  - Gifu Prefectural General Medical Center, Gifu
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Hirosaki University Hospital, Hirosaki-shi
  - Hiroshima University Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - Tomakomai City Hospital, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center, Hyōgo
  - Tokai University Hospital, Isehara
  - National Hospital Organization Kanazawa Medical Center, Ishikawa
  - Public Central Hospital of Matto Ishikawa, Ishikawa
  - Teikyo University Hospital, Itabashi Ku
  - Central Clinic, Kagoshima
  - Fukuoka Tokushukai Hospital, Kasuga-shi
  - Sekishinkai Second Kawasaki Saiwai Clinic, Kawasaki-shi
  - Kokura Memorial Hospital, Kitakyushu-shi
  - Kumamoto University Hospital, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Seikokai Omi Medical Center, Kusatsu-shi
  - Kyoto University Hospital, Kyoto
  - Ehime Prefectural Central Hospital, Matsuyama
  - Seijunkai Mito Hospital, Mito
  - Miyazaki Medical Association Hospital, Miyazaki
  - Miyakonojo Medical Association Hospital, Miyazaki
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - Saiseikai Narashino Hospital, Narashino-shi
  - Miwa Heart Clinic, Nishi-Tokyo-shi
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Okayama University Hospital, Okayama
  - Naha City Hospital, Okinawa
  - Watanabeigakukai Sakurabashi Watanabe Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Police Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Kindai University Hospital, Osaka Sayama Shi
  - Kitasato University Hospital, Sagamihara
  - Iwatsuki Minami Hospital, Saitama-shi
  - Matsuda Hospital, Sapporo
  - Sanseikai Miyanomori Memorial Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Showa University Hospital, Shinagawa City
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Japanese Red Cross Takatsuki Hospital, Takatsuki-shi
  - The Cardiovascular Institute Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Kenshinkai Minamino Cardiovascular Hospital, Tokyo
  - Ome Medical Center, Tokyo
  - Oji General Hospital, Tomakomai
  - Fujita Health University Hospital, Toyoake
  - Toyota Memorial Hospital, Toyota-shi
  - Uwajima City Hospital, Uwajima-shi
  - Yokohama Rosai Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Oita University Hospital, Yufu
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Lithuania (7):
  - Klinikiniai sprendimai JSC, Kaunas
  - Saules Seimos Medicinos Centras, JSC, Kaunas
  - Kaunas Clinical Hospital, Public Institution, Kaunas
  - Klaipeda Seamen's Hospital, Public Institution, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
  - Inlita, JSC, Vilnius
  - Inmedica, JSC, Vilnius
- Malaysia (8):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital University Sains Malaysia, Kota Bharu
  - Queen Elizabeth II Hospital, Kota Kinabalu
  - Institut Jantung Negara, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Universiti Teknologi Mara, Selayang Baru Utara
  - Hospital Seri Manjung, Seri Manjung
  - Hospital Taiping, Taiping
- Netherlands (23):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - ZGT Cardioresearch, Almelo
  - Meander Medisch Centrum, Amersfoort
  - VUMC Amsterdam, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - Atrium Med.Centrum Heerlen - Afd.Interne - INT, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Alrijne Ziekenhuis Leiden ; Cardiology, Leiderdorp
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Radboudumc, Nijmegen
  - Sint Franciscus Gasthuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - D & A Research, Sneek
  - ETZ Elisabeth, Tilburg
  - Maxima Medisch Centrum, Veldhoven
  - Gelre Ziekenhuizen Zutphen, Zutphen
- New Zealand (10):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - University of Otago, Christchurch
  - Dunedin Public Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Hawkes Bay Hospital, Hastings
  - Taranaki Base Hospital, New Plymouth
  - Middlemore Hospital, Otahuhu
  - Rotorua Hospital, Rotorua
  - Tauranga Hospital, Tauranga
- Philippines (9):
  - Silang Specialists Medical Center, Cavite
  - Perpetual Succour Hospital, Cebu City
  - Central Lab Diabetes Wellness, Heart and Kidneys, Inc, Davao City
  - Davao Doctors Hospital, Davao City
  - St.Paul's Hospital-Iloilo, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - St. Luke's Medical Center, Manila
  - GreenCity Medical Center, San Fernando City
  - Cardinal Santos Medical Center, San Juan City
- Poland (60):
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
  - IN VIVO Sp. z o.o, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne Intercor Sp z o o, Bydgoszcz
  - Centrum Medyczne PRATIA Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Pratia Chojnice, Chojnice
  - DIAB SERWIS Popenda Sp. Jawna Specjalistyczna Przychodnia Lekarska, Chorzów
  - M2M Badania Kliniczne, Chorzów
  - Centrum Medyczne MBB-MED, Chrzanów
  - NZOZ Twoje Zdrowie El, Elblag
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - Private Practice - Dr. Krzysztof Cymerman, Gdynia
  - NZOZ Procordis Pawel Miekus, Gdynia
  - MCBK Iwona Czajkowska Anna Podrazka Szczepaniak S C, Grodzisk Mazowiecki
  - Centrum Medyczne Pratia Jelenia Gora, Jelenia Góra
  - Centrum Medyczne Pratia Katowice, Katowice
  - Clinical Medical Research Sp. z o.o., Katowice
  - Silmedic sp. z o.o, Katowice
  - Kardio Klinika Brynow, Katowice
  - Niepubliczny Zaklad Opieki Zdrowotnej, Katowice
  - Specjalistyczna Poradnia Kardiologiczna i Nadcisnienia Tetniczego, Kielce
  - Ewa Mirek-Bryniarska Specjalistyczna Praktyka Lekarska, Krakow
  - Centrum Medyczne Linden, Krakow
  - Centrum Medyczne Zdrowa J Trebacz W Zajdel s j, Krakow
  - Krakowskie Centrum Medyczne Sp z o o NZOZ, Krakow
  - Odzial Kardiologii i Chorob Wewnetrznych Szpital Specjalistyczny im. Ludwika Rydygiera, Krakow
  - B.Miklaszewicz&D.Dabrowski CARDIMED Spolka Jawna, Legnica
  - SANTA FAMILIA Centrum Badan Profilaktyki i Leczenia, Lodz
  - Centrum Medyczne Med Gastr, Lodz
  - Centrum Medyczne AMED oddzial w Lodzi, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - NZOZ ALL-MED Centrum Medyczne Specjalistyczne Gabinety Lekarskie, Lodz
  - Indywidualna Specjalistyczna Praktyka Lekarska, Lodz
  - Lowickie Centrum Kardiologii, Lowicz
  - 1 Wojskowy Szpital Kliniczny Z Poliklinika SPZOZ W Lublinie, Lublin
  - KO MED Centra Kliniczne LUBLIN, Lublin
  - ETG Lublin, Lublin
  - FutureMeds Olsztyn, Olsztyn
  - Ostrowieckie Centrum Medyczne Spolka Cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski
  - Medicome Sp. Z O.O., Oświęcim
  - NZOZ Heureka, Piaseczno
  - Med-Polonia Sp. z o.o., Poznan
  - NZOZ NEURO KARD Ilkowski i Partnerzy Sp Partnerska Lekarzy, Poznan
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Janusz Spyra Specjalistyczna Praktyka Lekarska, Ruda Śląska
  - Centrum Medyczne Medyk, Rzeszów
  - ETG Siedlce, Siedlce
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej w Siedlcach, Siedlce
  - Centrum Medyczne Ogrodowa sp. z o.o., Skierniewice
  - FutureMeds Warszawa Centrum, Warsaw
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
  - ETG Warszawa, Warsaw
  - FutureMeds Targowek, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika SP ZOZ, Wroclaw
  - NZOZ Zdrowie s c Agnieszka i Donald Drozdz, Wroclaw
  - CM Sedimed Wroclaw, Wroclaw
  - ETG Zamosc, Zamość
  - Velocity Zamosc, Zamość
  - Centrum Medyczne Serafin med, Żarów
- Portugal (9):
  - Uls Coimbra - Hosp. Univ. Coimbra, Coimbra
  - Centro Hospitalar Cova da Beira, EPE - Hospital Pêro da Covilhã, Covilha
  - Hospital Distrital Fig Da Foz Gala, Figueira da Foz Municipality
  - Centro Hospitalar de Lisboa Norte Hospital Santa Maria, Lisbon
  - Centro Hospitalar Lisboa Ocidental - Hospital São Fracisco Xavier, Lisbon
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E, Santa Maria da Feira
  - Largo da Igreja Velha Edifício CCA, Torres Novas
  - Centro Hospitalar de Vila Nova de Gaia Espinho E P E, Vila Nova de Gaia
  - Centro Hospitalar de Trás os Montes e Alto Douro- Vila Real, Vila Real
- Romania (19):
  - CMI Cardiologie Dr. Calin Pop, Baia Mare
  - Centrul Medical Unirea SRL, Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulator NEOMED, Brasov
  - Spitalul Judetean de Urgenta Braila, Brăila
  - Clinica Medicala Data Plus SRL, Bucharest
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu si Medicina Preventiva, Bucharest
  - S C Delta Health Care S R L, Bucharest
  - Institutul de urgenta pentru Boli Cardiovasculare Prof. Dr. C.C. Iliescu, Bucharest
  - Spitalul Clinic de Urologie Prof. Dr. Theodor Burghele, Bucharest
  - Spitalul Angiocare SRL, Cluj-Napoca
  - Institutul de Boli Cardiovasculare Iasi, Iași
  - Cardiomed SRL, Iași
  - Spitalul Clinic Judetean de Urgenta Oradea, Oradea
  - SAL MED Pitesti, Piteşti
  - Spitalul Clinic Judetean Sibiu, Sibiu
  - Cabinet Medical Cardiologie Cojocariu Titel Razvan, Suceava
  - Cmi Dr Podoleanu Cristian, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Tg. Mures
  - Clinica Medicaliss, Timișoara
- Serbia (13):
  - Institute for Cardiovascular diseases Dedinje, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Clinical Center Bezanijska kosa, Belgrade
  - University Clinical Hospital Center Dr Dragisa Misovic- Dedi, Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - Clinical Center of Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - General Hospital Pancevo, Pančevo
  - General Hospital Smederevo, Smederevo
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
  - General Hospital Uzice, Užice
  - Health Center Zajecar, Zaječar
- Singapore (2):
  - National Heart Centre (NHC) Singapore, Singapore
  - Singapore General Hospital, Singapore
- Slovakia (22):
  - Alian s.r.o., Bardejov
  - Thyreomedical s r o, Bardejov
  - Cardioconsult s.r.o., Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
  - Kardiovaskularne centrum, s.r.o., Bratislava
  - Narodny ustav srdcovych a cievnych chorob, Bratislava
  - Veria, s.r.o Kardiologicka ambulancia, Bratislava
  - Nemocnica s poliklinikou Brezno, Brezno
  - KARDIO-ONKOLOGIA s.r.o. Kardiologicka ambulancia, Dolný Kubín
  - Východoslovenský Ústav Srdcových A Cievnych Chorôb, A.S., Košice
  - Cardio D&R, s.r.o., Košice
  - Kardiologicka ambulancia Medicalgroup s.r.o., Košice
  - IN-DIA s.r.o., Lučenec
  - Kardio 1 S.R.O., Lučenec
  - Kardiomed, S.R.O., Lučenec
  - Kardiologicka ambulancia MEDI M&M s.r.o., Moldava nad Bodvou
  - Fakultna nemocnica Nitra, Nitra
  - Cardioinvest s.r.o., Nové Zámky
  - Medispol s.r.o Interna a kardiologicka ambulancia, Prešov
  - Fakultna nemocnica s poliklinikou J.A. Reimana Presov, Prešov
  - Interna SK s.r.o., Svidník
  - MEDIVASA s.r.o., Žilina
- South Africa (10):
  - Tread Research, Cape Town
  - Johese Clinical Research, Centurion
  - Garda, RA, Johannesburg
  - DJW Research, Krugersdorp
  - Clinical Research Unit, University of Pretoria, Pretoria
  - Into Research, Pretoria
  - Dr J.M. Engelbrecht Trial Site, Somerset West
  - Helderberg Research Institute, Somerset West
  - Mediclinic Victoria Hospital, Tongaat
  - Clinical Projects Research SA (PTY) LTD, Worcester
- South Korea (32):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Dong-A University Hospital, Busan
  - Dankook University Hospital, Cheonan-si
  - Chungbuk National University Hospital, Cheongju-si
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Hanyang University Guri Hospital, Guri-si
  - Chonnam National University Hospital, Gwangju
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju Special
  - Chungnam National University Hospital, Sejong-si
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Kyung Hee University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - WonJu Severance Christian Hospital, Wŏnju
  - Yongin Severance Hospital, Yongin-si
- Spain (15):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Del Mar, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. de Bellvitge, Barcelona
  - Hosp. Univ. Virgen de La Arrixaca, El Palmar
  - Hosp. Univ. Arnau de Vilanova de Lleida, Lleida
  - Hosp. Virgen de La Luz, Madrid
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. de Manises, Manises
  - Hosp Virgen de La Victoria, Málaga
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (12):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Mackay Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan
- Turkey (Türkiye) (9):
  - Afyon Kocatepe University Medical Faculty, Afyonkarahisar
  - Turkiye Yuksek Ihtisas Training and Research Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Marmara University Pendik Training Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Erciyes University Medical Faculty, Kayseri
  - Mersin University Medical Faculty, Mersin
  - Mersin University Medical Faculty Hospital, Mersin
  - Ondokuz Mayis University, Samsun
- United Kingdom (12):
  - Bristol Royal Infirmary, Bristol
  - Golden Jubilee National Hospital, Clydebank
  - Dorset County Hospital, Dorchester
  - Royal Devon and Exeter Hospital(Wonford), Exeter
  - Wycombe Hospital, High Wycombe
  - Lincoln County Hospital, Lincoln
  - Barts Hospital, London
  - Northern General Hospital, Sheffield
  - Lister Hospital, Stevenage
  - Royal Cornwall Hospital, Truro
  - Wrightington Hospital,Wrightington, Wigan and Leigh NHS Trus, Wigan
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Jain SS, Mahaffey KW, Pieper KS, Shimizu W, Potpara T, Ruff CT, Kamel H, Lewis BS, Cornel JH, Kowey PR, Horrow J, Strony J, Plotnikov AN, Li D, Weng S, Donahue J, Gibson CM, Steg PG, Mehran R, Weitz JI, Johnston SC, Hankey GJ, Harrington RA, Lam CSP; LIBREXIA AF Trial Investigators and Committees. Milvexian vs apixaban for stroke prevention in atrial fibrillation: The LIBREXIA atrial fibrillation trial rationale and design. Am Heart J. 2024 Nov;277:145-158. doi: 10.1016/j.ahj.2024.08.011. Epub 2024 Aug 29. PMID 39214801